CLINICAL TRIAL: NCT05830903
Title: Develop a Novel Occupational Training Program for Schizophrenia Patients Based on Virtual Reality Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201904105RINB
Record Dates: First submitted 2019-07-04; First posted 2023-04-26 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia; Cognitive Impairment
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mild ED/NS (Experimental): 10 patients with mild or none executive function impairment and mild or none negative symptoms.
  Interventions: Behavioral: VR-assisted occupational training
- Mild ED/Severe NS (Experimental): 10 patients with mild or none executive function impairment and severe or moderate negative symptoms.
  Interventions: Behavioral: VR-assisted occupational training
- Severe ED/Mild NS (Experimental): 10 patients with severe or moderate executive function impairment and mild or none negative symptoms.
  Interventions: Behavioral: VR-assisted occupational training
- Severe ED/NS (Experimental): 10 patients with severe or moderate executive function impairment and severe or moderate negative symptoms.
  Interventions: Behavioral: VR-assisted occupational training

INTERVENTIONS:
Behavioral: VR-assisted occupational training — VR-assisted occupational training

SUMMARY:
Establish a novel vocational training program and test its validity in a pilot study.

DETAILED DESCRIPTION:
40 schizophrenia patients will be recruited to join the virtual reality based vocational training program, the training effect will be compared by interview skills and problem solving before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of schizophrenia based on the Diagnostic and Statistical Manual of Mental Disorders -5th version
* Aged between 20 and 55 years.
* Motivated to have a job.
* Having a full-scale IQ > 70 on the Wechsler Adult Intelligence Scale-version IV.
* Having a PANSS positive scale < 70, indicating a stable condition during the illness course.

Exclusion Criteria:

* Comorbid with other major psychiatric disorders (i.e., bipolar disorders) or neurological diseases.
* Substance abuse within one year.
* Visual impairment and/or hearing impairment that would preclude participation in the VR-based training program.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical ratings of schizophrenia symptoms | 8 weeks
  The Positive and Negative Syndrome Scale (PANSS) is a 30-item rating scale completed by trained research staff. Scores for positive, negative, cognitive disorganization, emotional discomfort, and hostility/excitement symptoms were derived from factor-derived scoring published.
  * There are 30 different symptoms rated from 1 to 7 (total score of 210). Higher the score, worse the symptoms
vocational skills | 8 weeks
  Job interview role-play performance will be scored across nine domains: conveying oneself as a hard worker, sounding easy to work with, conveying that one behaves professionally, negotiation skills (requesting one day off), sharing things in a positive way, sounding honest, sounding interested in the position, comfort level, and establishing rapport
global improvement | 8 weeks
  Clinical Global Impression Improvement scale (CGI-I) rating scales are commonly used measures of symptom severity, treatment response and the efficacy in treatment studies of patients with mental disorders. It is a 7-point scale that require clinician to assess how much the patient's illness has improved or worsened relative to baseline. "1" meaning very much improved, "7" meaning very much worsen.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ling Chien, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan